CLINICAL TRIAL: NCT02476955
Title: An Open-label Phase 1b Study of ARQ 092 in Combination With Other Antineoplastic Agents in Subjects With Selected Solid Tumors
Brief Title: Open-label Phase 1b Study of ARQ 092 in Combination With Anastrozole
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: ArQule, Inc., a subsidiary of Merck Sharp & Dohme LLC, a subsidiary of Merck & Co., Inc. (Rahway, NJ USA) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7075-001; ARQ 092-102 (Other: ArQule Study ID)
Record Dates: First submitted 2015-06-10; First posted 2015-06-22 (Estimated); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Solid Tumors; Ovarian Cancer; Endometrial Cancer
Keywords: ARQ 092; Carboplatin; Paclitaxel; AKT inhibitor in combination therapy; Targeted therapy; Molecular therapy; Tyrosine kinase inhibitor (TKI); Receptor tyrosine kinase (RTK); Biomarkers; Phase 1 - Phase I; Solid tumors; Metastatic solid tumors; Recurrent solid tumors; Ovarian cancer; Endometrial cancer; Cervical cancer; Triple-negative breast cancer; AKT kinases; AKT pathway; AKT signaling; AKT inhibitor; AKT pan inhibitor; Chemotherapy; PI3K/AKT/mTOR signaling pathway; AKT1; AKT2; AKT3; Phase I Clinical Trial; Clinical oncology; Tumor; AKT1 inhibitor; AKT2 inhibitor; AKT3 inhibitor; AKT1 mutation; AKT2 mutation; AKT3 mutation; AKT1 amplification; AKT2 amplification; AKT3 amplification; Anastrozole; Estrogen receptor positive; PIK3CA mutation
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms; Uterine Cervical Neoplasms; Triple Negative Breast Neoplasms; Neoplasms | interventions — Miransertib; Carboplatin; Paclitaxel; Albumin-Bound Paclitaxel; Anastrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ARQ 092 + anastrozole (Experimental): ARQ 092 will be administered orally at 150 milligrams (mg) every day (QD), 5 days on/9 days off of a 28 day cycle in combination with anastrozole which will be administered orally at 1 mg QD continuously. The combination treatment will continue until progression of disease (clinical or radiological), unacceptable toxicity, or another of the discontinuation criteria is documented.
  Interventions: Drug: ARQ 092 + carboplatin + paclitaxel (Closed); Drug: ARQ 092 + paclitaxel (Closed); Drug: ARQ 092 + anastrozole

INTERVENTIONS:
Drug: ARQ 092 + carboplatin + paclitaxel (Closed) — Subjects will receive ARQ 092 orally at dose levels specified for their respective dose cohorts plus carboplatin (AUC6, intravenously, Day 1) plus paclitaxel (175 mg/m2, intravenously, Day 1) on a 21-day schedule.
  Other Names: cis-Diammine; Paraplatin; Taxol; Abraxane
Drug: ARQ 092 + paclitaxel (Closed) — ARQ 092 will be administered orally at 200 mg twice a day (BID) weekly (Cohort 1P) of a 28-day cycle in combination with an intravenous (IV) infusion of paclitaxel (80 mg/m2). ARQ 092 will be administered once a week on Day 1, Day 8, Day 15, and Day 22 of each 28-day cycle; paclitaxel will be administered once a week on Day 1, Day 8, and Day 15 for three consecutive weeks followed by one week off of each 28-day cycle.
  Other Names: Taxol; Abraxane
Drug: ARQ 092 + anastrozole — ARQ 092 will be administered orally at 150 mg QD, 5 days on/9 days of a 28 day cycle in combination with anastrozole which will be administered orally at 1 mg QD continuously.
  Other Names: Arimidex

SUMMARY:
An Open-label Phase 1b Study of ARQ 092 in Combination with other Antineoplastic Agents in Subjects with Selected Solid Tumors

DETAILED DESCRIPTION:
This is an open-label Phase 1b, dose escalation study of oral ARQ 092 administered in combination with carboplatin plus paclitaxel (Carboplatin Plus Paclitaxel Arm) or in combination with paclitaxel alone (Paclitaxel Arm), in subjects with advanced, inoperable metastatic and/or recurrent solid tumors, or in combination with anastrozole (Anastrozole Arm) in subjects with ovarian or endometrial cancer.

Enrollment in the Carboplatin plus Paclitaxel Arm and Paclitaxel Alone Arm is now closed. Enrollment in the Expansion Cohort for the Anastrozole Arm continues for patients with Endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent form
2. 18 years of age or older
3. Histologically or cytologically confirmed locally advanced, inoperable, or metastatic tumors:

   * Subjects with endometrial cancer with:

     * Documented/locally determined AKT1, PIK3CA, or PIK3R1 mutations with or without PTEN deficiency
     * ER+ status
4. Female subjects of child-bearing potential must have a negative serum or urine pregnancy test within 72 hours prior to administration of the first dose of study drug. "Women of childbearing potential" is defined as sexually mature women who have not undergone hysterectomy and/or bilateral oophorectomy, or who have not been naturally postmenopausal for at least 12 consecutive months prior to administration of the first dose of the study drug.
5. Measurable or evaluable disease
6. Subjects must agree to provide requested amount of archival and/or fresh tissue biopsy samples at baseline for mutational analysis by the Sponsor's central laboratory.
7. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
8. Life expectancy ≥ 12 weeks
9. Failure to respond to or refractory to approved/standard therapy; or for whom standard therapy does not exist, or is not tolerable; or for whom approved/standard therapy is not considered to be sufficient or appropriate by the Investigator.
10. Adequate organ function as indicated by the following laboratory values. All laboratory tests must be obtained within 7 days prior to the first dose of study treatment:

    * Hematological

      - Absolute neutrophil count (ANC) ≥ 1.0 x 109/L

      - Platelet count (Plt) ≥ 100 x 109/L

      - Hemoglobin (Hb) ≥ 8 g/dL
    * Renal

      * Serum creatinine ≤ 1.5 x upper limit of normal (ULN) or
      * Calculated creatinine clearance ≥ 60 mL/min /1.73 m2 for subjects with serum creatinine levels > 1.5 x institutional ULN
    * Hepatic

      * Total bilirubin ≤ 1.5 x ULN or
      * Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 x ULN
      * AST and ALT ≤ 3 x ULN or ≤ 5 x ULN for subjects with known liver metastases
    * Metabolic - Glycated hemoglobin (HbA1c) ≤ 8%
11. If a subject is currently receiving bisphosphonates or denosumab, the subject must have received the bisphosphonates or denosumab for at least four weeks before starting study treatment. Initiation of bisphosphonates or denosumab during the study may be allowed provided the subject completes the first cycle of treatment without any DLT and the Investigator rules out tumor progression.
12. Male or female subjects of child-bearing potential must agree to use double-barrier contraceptive measures, oral contraception, or avoidance of intercourse during and after the study (3 months after the last dose of ARQ 092 or anastrozole, whichever is longer)

Exclusion Criteria:

1. Anti-cancer therapy, such as chemotherapy, immunotherapy, targeted and hormonal/endocrine therapy, or investigational agents within five half-lives or two weeks (whichever is shorter) for oral drugs, five half-lives or four weeks (whichever is shorter) for intravenous drugs, and six weeks for nitrosoureas, mitomycin C, or bevacizumab prior to administration of the first dose of study drug

   * To be eligible for study treatment, toxicity from prior treatment must recover to Grade ≤ 1, except for alopecia
   * Concurrent systemic high-dose corticosteroids when used intermittently in an antiemetic regimen for central nervous system (CNS) metastases management or as a part of the premedication regimen are allowed
   * Prior hormonal therapy (including, but not limited to, tamoxifen, megestrol acetate, fulvestrant, and GnRH analogs) for the treatment of recurrent/advanced endometrial cancer are not allowed
2. Radiation therapy within four weeks prior to administration of the first dose of study drug

   • To be eligible for study treatment, radiation therapy-related toxicity must recover to Grade ≤ 1 prior to administration of the first dose of study drug. Concurrent palliative radiotherapy for local pain-control may be allowed, provided the subject does not meet criteria of progressive disease and treated lesions will not be included in the target/non-target lesion assessment.
3. Major surgical procedure within four weeks prior to administration of the first dose of study drug

   • To be eligible for study treatment, all surgical wounds must be fully healed and any surgery-related adverse events (AE) must recover to Grade ≤ 1
4. Previous treatment with AKT inhibitors (e.g., MK-2206, GSK2141795, AZD5363)
5. Contraindications to treatment with anastrozole defined by the Investigator based on institutional Standard of Care (SOC), scientific evidence, expert medical judgment, or published literature
6. History of allergic reaction attributed to compound(s) of similar chemical or biologic composition as ARQ 092 or anastrozole
7. Unable or unwilling to swallow ARQ 092 or anastrozole
8. Known active Central Nervous System (CNS) metastases and/or carcinomatous meningitis

   • To be eligible for the study treatment, subjects must have stable disease ≥ 3 months, confirmed by magnetic resonance imaging (MRI) or computed tomography (CT) scan, and have CNS metastases well controlled by low-dose steroids, anti-epileptics, or other symptom-relieving medications
9. History of myocardial infarction (MI) or congestive heart failure defined as Class II to IV per the New York Heart Association (NYHA) classification within 6 months of the first dose of ARQ 092 (MI that occurred > 6 months prior to the first dose of ARQ 092 will be permitted)
10. History of Type 1 or 2 diabetes mellitus requiring regular medication (other than oral hypoglycemic agents including metformin) or fasting glucose ≥ 160 mg/dL
11. Significant gastrointestinal disorder(s), that could in the opinion of the Investigator, interfere with the absorption, metabolism, or excretion of ARQ 092 (e.g., Crohn's disease, ulcerative colitis, extensive gastric resection)
12. Previous malignancy within 2 years of the first dose of study drugs, except tumors totally resected and/or not requiring therapy
13. Concurrent uncontrolled illness not related to cancer, including but not limited to:

    • Ongoing or active infection, including human immunodeficiency virus (HIV), hepatitis B (HBV) (hepatitis B surface antigen [HBsAg] positive; subjects with documented laboratory evidence of HBV clearance may be enrolled) or hepatitis C (HCV) (positive HCV antibody), or bleeding
14. Psychiatric illness, substance abuse, and/or social situation that would limit compliance with study requirements
15. Blood transfusion within 5 days of the blood draw being used to confirm eligibility
16. Pregnant or breastfeeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-06-09 (Actual); Primary Completion 2019-05-07 (Actual); Study Completion 2019-05-07 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events (TEAEs) as assessed by the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 | Assessed at each scheduled visit up to treatment discontinuation + 30 days with an estimated treatment duration of 3 to 24 weeks
  The incidence of adverse events will be assessed as a measure of the safety and tolerability profile of ARQ 092
Overall Response Rate (ORR) based on central review of tumor measurement using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 | Baseline and every 2 cycles (8 weeks) after the first dose of ARQ 092 during the first 6 cycles (24 weeks) of treatment, and every 3 cycles (12 weeks) thereafter or as clinically indicated, and at the End of Treatment.
  ORR will be assessed as a measure of efficacy
Progression Free Survival (PFS) based on central review of tumor measurement using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 | Baseline and every 2 cycles (8 weeks) after the first dose of ARQ 092 during the first 6 cycles (24 weeks) of treatment, and every 3 cycles (12 weeks) thereafter or as clinically indicated, and at the End of Treatment.
  PFS will be assessed as a measure of efficacy
Duration of Response (DoR) based on central review of tumor measurement | Baseline and every 2 cycles (8 weeks) after the first dose of ARQ 092 during the first 6 cycles (24 weeks) of treatment, and every 3 cycles (12 weeks) thereafter or as clinically indicated, and at the End of Treatment.
  DoR will be assessed as a measure of efficacy

SECONDARY OUTCOMES:
Peak plasma concentration (Cmax) | During Cycle 1, Day 1 and Cycle 2, Day 1 of treatment (t=0, 2, 4, 6, 8, 10, 12 hours post ARQ 092 dose). And at Cycle 1, Day 8, Day 15, and Day 22 (t = pre-dose ARQ 092 dose).
Area under the plasma concentration vs. time curve (AUC) | During Cycle 1, Day 1 and Cycle 2, Day 1 of treatment (t=0, 2, 4, 6, 8, 10, 12 hours post ARQ 092 dose). And at Cycle 1, Day 8, Day 15, and Day 22 (t = pre-dose ARQ 092 dose).
Half-life of ARQ 092 | During Cycle 1, Day 1 and Cycle 2, Day 1 of treatment (t=0, 2, 4, 6, 8, 10, 12 hours post ARQ 092 dose). And at Cycle 1, Day 8, Day 15, and Day 22 (t = pre-dose ARQ 092 dose).

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Grand Rapids, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - MD Anderson Cancer Center, Houston, Texas
  - San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php